CLINICAL TRIAL: NCT00218582
Title: Effectiveness of Self-Help for Dually-Diagnosed Persons
Brief Title: Effectiveness of Self-Help for Dually-Diagnosed Persons - 1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: National Development and Research Institutes, Inc. (Other)
Responsible Party: Stephen Magura, Western Michigan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-15912-1; R01-15912-1
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-10

CONDITIONS: Dual Diagnosis; Substance-Related Disorders; Mental Disorders
Keywords: 12 step groups; self help; psychiatric day treatment; co-occurring disorders; dual diagnosis
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dual focus 12 step mutual aid groups for persons with co-occurring disorders (psychiatric and substance use disorders), provided within the context of standard psychiatric day treatment
  Interventions: Behavioral: Double Trouble in Recovery
- 2 (Active Comparator): Standard psychiatric day treatment
  Interventions: Behavioral: Standard psychiatric day treatment

INTERVENTIONS:
Behavioral: Double Trouble in Recovery — Dual focus 12 step mutual aid groups for persons with co-occurring disorders (psychiatric and substance use disorders), provided within the context of standard psychiatric day treatment
  Arms: 1
Behavioral: Standard psychiatric day treatment — Individual counseling, groups, medication
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effectiveness of adding dual focus 12-step self-help groups to standard treatment to improve behavioral outcomes for patients dually diagnosed with substance abuse and psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

Admission to psychiatric day treatment program 18-64 years old

Exclusion Criteria:

Did not understand or speak English, appeared intoxicated on drugs or alcohol, carried a diagnosis of mental retardation, were deemed actively psychotic by the clinic's intake coordinator, appeared unable to understand and give informed consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2003-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
drug/alcohol use | past 90 days

SECONDARY OUTCOMES:
psychiatric medication adherence | recent
traditional 12 step meeting attendance | past 90 days
psychiatric symptoms | recent
program retention | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Magura, Ph.D., Principal Investigator — National Development and Research Institutes, Inc.
Locations (1):
- Albert Einstein Dept of Psychiatry, The Bronx, New York, United States

REFERENCES:
- [Result] Magura S, Rosenblum A, Villano CL, Vogel HS, Fong C, Betzler T. Dual-focus mutual aid for co-occurring disorders: a quasi-experimental outcome evaluation study. Am J Drug Alcohol Abuse. 2008;34(1):61-74. doi: 10.1080/00952990701764623. PMID 18161644